CLINICAL TRIAL: NCT01781195
Title: Effect of Delayed CNI-based Immunosuppression With Advagraf on Liver Function After MELD-based Liver Transplantation
Brief Title: Delayed CNI-based Immunosuppression With Advagraf After MELD-based Liver Transplantation
Acronym: IMUTECT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Principal Investigator, Peter Schemmer, professor, Heidelberg University
Other Study IDs: IMUTECT2013-01
Record Dates: First submitted 2013-01-29; First posted 2013-01-31 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Liver Graft Dysfunction
Keywords: Advagraf; MELD-score; Na-MELD-score; liver function; LiMAx-test; infection rate; HLA-DR status; immunostatus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood: HLA-DR status
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Advagraf-based immunosuppression: 50 patients after liver transplantation (25 with a MELD-score ≤20 and 25 patients with a MELD-score >20) under CNI-based immunosuppression with Advagraf

SUMMARY:
Prolonged-release low-dose Advagraf should better protect from CNI-side effects compared to standard immunosuppressive regiments while the rate of rejection is not increased and thus graft function is well maintained. We hypothesize that especially in high-MELD (MELD-score >20) recipients who have a decreased immune competence the prolonged-release low-dose Advagraf concept would better protect from side effects of immunosuppression (i.e. infection). Nevertheless, we assume that also patients with a MELD-score ≤20 will benefit from this concept in regard to lower infection rates and less side effects of immunosuppression.

DETAILED DESCRIPTION:
The MELD-score (model of end stage liver disease) was designed to estimate the prognosis after TIPS (transjugular intrahepatic porto-systemic shunt). Nowadays it is the key-score for patients awaiting a liver graft and consists of serum-creatinine, serum-bilirubine and the INR-ratio with values between 6-40. The MELD-based liver allocation follows the sickest patient first strategy which significantly decreased outcome after liver transplantation (LTx) in Germany. There is evidence that the immune competence of very sick patients is decreased. Monocytic HLA-DR status is a marker for the function of the immune system. A reduced monocytic HLA-DR expression is indicative for a suppressed immune system.

Blood levels of Advagraf are slowly increased during the first week until the aimed tacrolimus trough levels are reached. Since therapeutic tacrolimus trough levels are reached not before the end of the first week after transplantation this is a concept for prolonged-release immunosuppression.

We assume, that high-MELD patients (MELD >20) undergoing LTx are immunosuppressed per se. Thus prolonged-release low-dose immunosuppression with Advagraf would decrease both- infection rate (CMV-reactivation, wound infection urinary tract infections, pneumonia, etc.) and side effects of immunosuppression. The immune capacity of patients will be determined by the measurement of monocytic HLA-DR status. To ensure that graft function is not impaired due to rejection episodes, liver function will be determined with the LiMAx-test, a routine procedure in our institution. After 13-C-Methacetin is given to the patient, it is metabolized to paracetamol and 13CO2 by the enzyme CYP1A2 which is localized in hepatocytes. The 13CO2/12CO2 ratio in the exhaled air correlates with liver function.

ELIGIBILITY:
Inclusion Criteria:

* age >18, <65
* first liver transplantation
* Immunosuppression with Advagraf, MMF, corticosteroid
* surgery and postoperative treatment at the department for general-, visceral- and transplantation surgery

Exclusion Criteria:

* missing informed consent
* re-transplantation
* acute infection: CMV (pp65 positive), pneumonia, urinary tract infection, wound infection, reactivation of Hepatitis B/C

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients with different MELD-scores/Na-MELD-scores undergoing liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-08 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
infection rate (CMV reactivation, wound infection, urinary tract infection, pneumonia) | 1-year follow-up per patient
  clinical visit: infection rate (CMV reactivation, wound infection, urinary tract infection, pneumonia)

SECONDARY OUTCOMES:
liver function (LiMAx) | one week
  LiMAx test before liver transplantation, and on postoperative days 1, 3, 7
HLA-DR status | one week
  HLA-DR status will be measured before liver transplantation and on postoperative days 3, 5, 7.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Schemmer, Prof., Principal Investigator — University Hospital Heidelberg
Locations (1):
- University Surgical Clinic, Heidelberg, Germany

REFERENCES:
- [Derived] Richter S, Polychronidis G, Gotthardt DN, Houben P, Giese T, Sander A, Dorr-Harim C, Diener MK, Schemmer P. Effect of delayed CNI-based immunosuppression with Advagraf(R) on liver function after MELD-based liver transplantation [IMUTECT]. BMC Surg. 2014 Sep 1;14:64. doi: 10.1186/1471-2482-14-64. PMID 25178675